CLINICAL TRIAL: NCT07123103
Title: A Dose Escalation and Expansion Study of XB371 Administered in Participants With Locally Advanced or Metastatic Solid Tumors
Brief Title: A Study of XB371 Administered in Participants With Locally Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XB371-101
Record Dates: First submitted 2025-08-08; First posted 2025-08-14 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Solid Tumors
Keywords: Advanced Solid Tumors; Metastatic Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose-escalation Cohorts (Experimental): Participants will receive escalating doses of XB371 every 3 weeks of a 21-day cycle (alternate schedules may be evaluated) until meeting the criteria for treatment discontinuation.
  Interventions: Drug: XB371
- Dose-expansion Cohorts: Part A (Experimental): Participants with Tumor Type 1 (tumor type will be selected based on available data) will be randomized to receive XB371 at one of two recommended dose levels (recommended dose [RD]-1 or RD-2) every 3 weeks of a 21-day cycle (alternate schedules may be evaluated) until meeting the criteria for treatment discontinuation.
  Interventions: Drug: XB371
- Dose-expansion Cohorts: Part B (Experimental): Participants with Tumor Type 2 (tumor type will be selected based on available data) will receive XB371 at the recommended dose level every 3 weeks of a 21-day cycle (alternate schedules may be evaluated) until meeting the criteria for treatment discontinuation.
  Interventions: Drug: XB371

INTERVENTIONS:
Drug: XB371 — Intravenous (IV) infusion.

SUMMARY:
The primary purpose of the study is to characterize the safety and tolerability of XB371. The dose-escalation cohorts and Part B of the expansion cohorts are non-randomized. Part A of the expansion cohorts is randomized.

ELIGIBILITY:
Key Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
* Minimum life expectancy of ≥ 12 weeks.
* Recurrent locally advanced or metastatic solid tumors.
* Adequate end organ and bone marrow function.

Key Exclusion Criteria:

* Primary brain tumors or known active brain metastases, leptomeningeal, or cranial epidural disease.
* History of interstitial lung disease (ILD) of any grade or history of organizing pneumonia.
* Has acute ocular infection, acute or chronic ulcerative/cicatricial condition of conjunctiva or cornea.
* Known history of immunodeficiency virus (HIV) unless specific criteria are met.
* Active infection with hepatitis C virus (HCV) defined as positive for HCV antibody.
* Major surgery within 4 weeks before the first dose of study treatment.
* Received radiation therapy within 2 weeks before the first dose of study treatment.
* Received prior systemic anticancer therapy including investigational agents within 4 weeks before the first dose of study treatment.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with a Dose-limiting Toxicity (DLT) | Up to the end of the first cycle (Up to Day 21 of a 21-day cycle)
Number of Participants with a Treatment-emergent Adverse Event (TEAE) | Up to approximately 7 months

SECONDARY OUTCOMES:
Area Under the Plasma Concentration-time Curve (AUC) of XB371, Total Antibody and Unconjugated Belotecan | Up to approximately 7 months
Maximum Observed Plasma Concentration (Cmax) of XB371, Total Antibody and Unconjugated Belotecan | Up to approximately 7 months
Time to Maximum Observed Plasma Concentration (Tmax) of XB371, Total Antibody and Unconjugated Belotecan | Up to approximately 7 months
Trough Observed Plasma Concentration (Ctrough) of XB371, Total Antibody and Unconjugated Belotecan | Up to approximately 7 months
Number of Participants with Antidrug Antibodies to XB371 | Up to approximately 7 months
Dose-escalation Cohorts Only: Recommended Dose(s) for Expansion | Through completion of dose-escalation (up to approximately 18 months)
Dose-expansion Cohorts Only: Objective Response Rate as Assessed by the Investigator per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) | Up to approximately 18 months
Dose-expansion Cohorts Only: Duration of Response as Assessed by the Investigator per RECIST v1.1 | Up to approximately 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Exelixis
Locations (5):
- United States (5):
  - Exelixis Clinical Site #5, Rogers, Arkansas
  - Exelixis Clinical Site #4, Orlando, Florida
  - Exelixis Clinical Site #3, Grand Rapids, Michigan
  - Exelixis Clinical Site #2, Huntersville, North Carolina
  - Exelixis Clinical Site #1, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No